CLINICAL TRIAL: NCT02993601
Title: Evaluation of the Safety and Feasibility of a New Peripheral Oedema Monitor for Home and Clinical Use for Heart Failure Patients, Using the Heartfelt-1 Device
Brief Title: Feasibility Study of a New Peripheral Oedema Monitor for Heart Failure
Status: Completed | Type: Observational
Sponsor: Heartfelt Technologies (Industry)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RBH01
Record Dates: First submitted 2016-12-05; First posted 2016-12-15 (Estimated); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure, Diastolic; Edema Brain; Decompensated Heartfailure
Keywords: Heart Failure; Edema; Oedema; Decompensated Heartfailure
MeSH Terms: conditions — Heart Failure, Diastolic; Brain Edema; Heart Failure; Edema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 20 outpatients with peripheral oedema: 20 outpatients with clinically detectable peripheral oedema for 1 set of measurements.
  Interventions: Device: Heartfelt-1; Device: Weighing scales; Other: Medical grading of oedema; Other: Baseline assessements; Device: Water displacement method; Device: Callipers measurements; Device: Measuring tape
- 20 cardiology controls: 20 outpatients with heart failure without clinically detectable peripheral oedema (control group) for 1 set of measurements.
  Interventions: Device: Heartfelt-1; Device: Weighing scales; Other: Medical grading of oedema; Other: Baseline assessements; Device: Water displacement method; Device: Callipers measurements; Device: Measuring tape
- 10 in-patients peripheral oedema: 10 in patients hospitalised as a result of heart failure and fluid congestion with peripheral oedema, those patients will have several sets of measurements taken over time to measure the reduction of peripheral oedema which is likely to show common features with the formation of peripheral oedema.
  Interventions: Device: Heartfelt-1; Device: Weighing scales; Other: Medical grading of oedema; Other: Baseline assessements; Device: Water displacement method; Device: Callipers measurements; Device: Measuring tape
- 30 control without cardiac conditions: less than 30 normal controls (healthy volunteers and patients without heart failure) in the age group 55 and above who agree to have images taken using the Heartfelt-1 device (not the whole set of measurements).
  Interventions: Device: Heartfelt-1

INTERVENTIONS:
Device: Heartfelt-1 — The patients will stand in front of the Heartfelt-1 in order for images to be captured and the volume of their lower legs measured.
  Other Names: HF-1
Device: Weighing scales — The patient will be asked to stand on standard medical weighing scales, to measure their weight.
  Groups: 10 in-patients peripheral oedema; 20 cardiology controls; 20 outpatients with peripheral oedema
Other: Medical grading of oedema — A member of the research team will assess the severity of the peripheral oedema on a scale of 1-5.
  Groups: 10 in-patients peripheral oedema; 20 cardiology controls; 20 outpatients with peripheral oedema
Other: Baseline assessements — At the point study participants are recruited, their age, sex, diagnosis, aetiology of heart failure, LVEF (Left ventricular ejection fraction), medical and device therapy, time since diagnosis, BNP (B-type Natriuretic Peptide), CRP (C-Reactive Protein), renal function (EGFR), Haemoglobin, albumin and urinalysis will be assessed unless recent (less that 6 months old) results are available. The number of Heart failure hospital admissions in the last 2 years, LACE score, co-morbidities will also be noted.
  Groups: 10 in-patients peripheral oedema; 20 cardiology controls; 20 outpatients with peripheral oedema
Device: Water displacement method — This will involve filling a gauge with lukewarm water (27-35oC +-2oC) up to the appropriate level. The appropriate level is determined by the water stabilising after some has flown out of the gauge into the waste bucket. Once the water level is stable the patient, who is sitting on a chair will be gently plunging the foot (naked) in the gauge until their foot is flat on the bottom on the gauge. The water flowing out of the gauge into the measuring bucket will be collected until the flow of water stops. Four small marks with non-toxic /non-permanent pen will be made on the lower leg of the patient to indicate where the water level was at. The water which has been collected in the measuring bucket will be weighted with precision scales to determine the volume of water displaced by the insertion of the foot. The patient's foot will then be dried.
  Groups: 10 in-patients peripheral oedema; 20 cardiology controls; 20 outpatients with peripheral oedema
Device: Callipers measurements — This will involve making 4 marks on one of the foot/lower leg (small cross) using non-toxic / non- permanent pen. The measurement will consist of making 6 measurements between those marks using callipers, and reporting the distance on a calibrated tape.
  Groups: 10 in-patients peripheral oedema; 20 cardiology controls; 20 outpatients with peripheral oedema
Device: Measuring tape — The measurements taken using a medical tape measure will involve the circumference of the ankle to be measured as well as the circumference at the level of the arch of the foot. The medical tape used will be a CE marked disposable medical measuring tape to minimise the risk of infection. The measurements will be done on both feet.
  Groups: 10 in-patients peripheral oedema; 20 cardiology controls; 20 outpatients with peripheral oedema

SUMMARY:
The study aims at assessing the usefulness of the Heartfelt1 device in patients suffering from heart failure, who have peripheral oedema. The device is non-contact and does not requires patient compliance to work. It gives an output reading of the patient's lower leg volume.

During the study, this measurement will be compared to clinical standard and gold standard measurements as well as clinical grading of peripheral oedema.

DETAILED DESCRIPTION:
The Heartfelt-1 device is a CE (Conformité Européenne = European Conformity) mark medical device used to measure biometric parameters of the foot and lower leg. The study aims at assessing the usefulness in patients suffering from heart failure, who have peripheral oedema. Models used for the measurements of foot and lower legs have not yet been validated for this group of patients, who are likely to have feet with abnormal surface contours and appearance secondary to oedema. Peripheral oedema can be a leading indicator of heart failure de-compensation which can lead to hospitalisation of patients, and therefore the device could be a useful clinical tool to monitor patients in their home. The Heartfelt-1 device has the ability to recognise the patient's feet (amongst an average size household setting), and trigger automatically the measurements when the feet are naked (for example as the patient goes in and out of bed). This makes the device an obvious choice for patients with compliance issues with current methods of monitoring (e.g. daily use of weighing scales) and treatment (e.g. diuretics) if it could be validated in this patient group.

The study has two general aims:

The first is to collect a time-series of data on inpatients with peripheral oedema caused by heart failure, as they receive intravenous or oral diuretic treatment to remove excess fluid and achieve optimal body weight and fluid balance. This data will be used both to determine the attainable resolution of foot biometric measurements on a patient as their fluid status changes, and also to further develop the algorithms used in the device and make them usable on a wide range of feet/lower legs which have been deformed by oedema. The data required for this study are images taken using the Heartfelt-1 device, as well as validation measurements such as the figure of eight using a medical grade tape measure, callipers, or the water displacement method using a volumetric gauge, at multiple time-points whilst the peripheral oedema reduces.

The second, on a second group of stable ambulatory (Heart Failure) HF patients with variable levels of oedema, is to evaluate the performance of the Heartfelt-1 device in determining foot biometric parameters one a wide range of patients at a single point in time. Patients with stable chronic heart failure will have their foot/lower legs measured by the Heartfelt-1 device, as well as standard medical measurement (figure of eight using a medical grade tape measure, callipers) and gold standard measurement (water displacement method using a gauge), as well as the patient's weight and a clinical grading of oedema. These will be compared and an estimate of the accuracy of the Heartfelt-1 device over this wider patient group can be extrapolated.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with admission for de-compensated heart failure requiring increase or initiation of diuretic therapy for fluid congestion.
* Patients attending cardiology outpatients at the Royal Brompton hospital with a diagnosis of heart failure and fluid retention.
* Cardiology patient without fluid retention (cardiology controls) Non-Cardiology patient without fluid retention (controls)

Exclusion Criteria:

* Patients unable to provide informed consent.
* Unstable arrhythmias in previous 48 hours
* Systolic BP<90mmHg or need for inotropic support
* Ulceration on lower limbs (below shin) - excluded from water displacement but could have image recording and calipers
* Inability to transfer from bed to chair
* Patients with broken skin or cellulitis will not have their foot volume measured using the water displacement equipment to reduce the risk of infection for the patient and other participants.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults able to give consent to take part in the study
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2017-06-13 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
Volume as measured by the Heartfelt-1 device | Within 3 months after patient recruitment or before the end of the study (whichever is soonest).

SECONDARY OUTCOMES:
Weight | Within 3 months after patient recruitment or before the end of the study (whichever is soonest).
  Patient weight on the day
Distance measurements | Within 3 months after patient recruitment or before the end of the study (whichever is soonest).
  Distance measurements on the foot / lower leg of the patient
Circumference and "figure of eight" | Within 3 months after patient recruitment or before the end of the study (whichever is soonest).
  Lower leg / foot circumference and "figure of eight" measurement
Volume of the lower leg/foot | Within 3 months after patient recruitment or before the end of the study (whichever is soonest).
  As measured using the water displacement method.
Medical grading of oedema | Within 3 months after patient recruitment or before the end of the study (whichever is soonest).
  Medical grading of peripheral oedema on a scale 1-5

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Lyon, BCh PhD FRCP, Principal Investigator — Royal Brompton and Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We are not planning to share individual participant data with other researchers.

REFERENCES:
- [Result] Chausiaux O, Williams G, Nieznanski M, Bagdu A, Downer P, Keyser M, Husheer S. Evaluation of the Accuracy of a Video and AI Solution to Measure Lower Leg and Foot Volume. Med Devices (Auckl). 2021 Apr 13;14:105-118. doi: 10.2147/MDER.S297713. eCollection 2021. PMID 33880069